CLINICAL TRIAL: NCT03506906
Title: The Debated Role of Sleep Studies in Patients Under Established Home Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WI_18-023
Record Dates: First submitted 2018-04-12; First posted 2018-04-24 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Hypoventilation Syndrome; Chronic Obstructive Pulmonary Disease; Obesity Hypoventilation Syndrome; Restrictive Lung Disease; Neuromuscular Diseases
Keywords: Chronic hypoventilation syndrome; Polysomnography; Transcutaneous Capnometry; Noninvasive Ventilation; home mechanical ventilation; Ventilator´s set-up
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Obesity Hypoventilation Syndrome; Neuromuscular Diseases | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional-approach (Active Comparator): The non-invasive ventilation therapy will be optimized according to routine tests (blood gas analysis, lung function, ventilator's built-in software analysis)
  Interventions: Diagnostic Test: Routine tests
- Sleep studies-based approach (Experimental): Additionally to the routine tests, the results of a nocturnal polysomnography and transcutaneous capnometry under the non-invasive ventilation therapy will be considered for the therapy optimization.
  Interventions: Diagnostic Test: Sleep studies under noninvasive ventilation therapy; Diagnostic Test: Routine tests

INTERVENTIONS:
Diagnostic Test: Sleep studies under noninvasive ventilation therapy — Polysomnography Transcutaneous capnography
  Arms: Sleep studies-based approach
Diagnostic Test: Routine tests — Spirometry, six minute walk test, blood gas analysis, questionnaires (Epworth sleepiness score, health related quality of life severe respiratory insufficiency questionnaire)

SUMMARY:
Patients suffering chronic hypercapnic respiratory insufficiency (e.g. in chronic obstructive pulmonary disease, obesity hypoventilation syndrome) benefit from home mechanical ventilation. These patients are complex; and the ventilator´s parameters should be set-up according to the underlying disease and particular patient's characteristics. The non-invasive ventilation therapy is mostly titrated while the patient is awake, hence Problems, such as Patient-Ventilator asynchrony, arising while sleeping on the ventilator therapy would remain undetected.

Sleep studies, such as polysomnography or polygraphy and transcutaneous carbon dioxide monitoring could be valuable tools to fine-tune the ventilator's settings. This could foster the ventilator´s effectivity and patient satisfaction, thus therapy's adherence. Nevertheless the sleep studies are expensive, time-consuming and not widely available.

The aim of this study is to learn the findings of sleep studies when they are performed on stable patients on home mechanical ventilation as part of their routine check-ups. In this context, it will be assessed whether the sleep studies' findings lead to a change (adjustment) of the ventilator´s therapy. Moreover, this study aims to investigate whether the absence of sleep studies would result in missing important events that require an adjustment of therapy. The results of this study could provide information that lead to a more standardized protocol of follow-up checks of patients on home mechanical ventilation in a cost-effective manner.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hypercapnic respiratory failure secondary to one or more identified condition(s) (chronic obstructive pulmonary disease, obesity hypoventilation syndrome, neuromuscular diseases, restrictive lung diseases)
* Home mechanical ventilation for ≥ 6 months
* Stable condition for ≥ 1 month

Exclusion Criteria:

* Previous adjustment of the noninvasive ventilation therapy under sleep studies in the last 6 months
* Current respiratory exacerbation
* Any current comorbidity decompensation
* Any medical or psychological condition impairing the patient's ability to provide informed consent
* Missing signed informed consent
* Total sleep time during polysomnography <180 min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-11-11 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
Adjustment of non-invasive ventilation | One day
  Each case will be evaluated separately by 2 investigators. One of them will be provided with the diurnal evaluations only (as routinely); the second investigator will additionally have access to the sleep studies. Each investigator will classify the case as one of the following labels (primary outcome):
  1. Non-invasive ventilation therapy optimization is not required (all ventilator's parameters should stay unchanged)
  2. Optimization of non-invasive ventilation therapy is required (one or more of the ventilator's parameters should be re-set, irrespective of the magnitude)

SECONDARY OUTCOMES:
Non-invasive ventilation compliance | 6 months
  The ventilator's optimization will be performed randomly according to the clinical-based approach or the sleep studies-based approach. In the next follow-up visit, both arms will be re-evaluated. The change in non-invasive ventilation therapy compliance will be explored based on the ventilator´s built-in software data.
Health-related quality of life: questionnaire | 6 months
  In the next follow-up visit, the health-related quality of life of both groups will be evaluated with the severe respiratory insufficiency questionnaire.
arterial level of carbon dioxide | 6 months
  In the next follow-up visit, the arterial level of carbon dioxide of both groups will be evaluated in the blood gas analysis

CONTACTS AND LOCATIONS:
Overall Officials: Winfried J Randerath, Prof. Dr., Principal Investigator — Krankenhaus Bethanien
Locations (1):
- Krankenhaus Bethanien, Solingen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No